CLINICAL TRIAL: NCT05666908
Title: High-flow Nasal Oxygenation Improves Blood Oxygen Saturation During Asphyxia During Pulmonary Surgery With Double-lumen Endotracheal Intubation: a Randomized Controlled Study
Brief Title: HFNO Improves Blood Oxygen Saturation During Asphyxia During Pulmonary Surgery With Double-lumen Endotracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20223357001
Record Dates: First submitted 2022-09-21; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-09

CONDITIONS: Lung Neoplasms; Pneumothorax
MeSH Terms: conditions — Lung Neoplasms; Pneumothorax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFNO group (Experimental): Direct guidance and positioning of DLT intubation with FOB visualization, using HFNO during intubation asphyxia.
  Interventions: Device: HFNO
- Control group (No Intervention): The DLT cannula was directly guided and positioned under FOB visualization, and no oxygen therapy equipment was used during intubation.

INTERVENTIONS:
Device: HFNO — After the patient's mask-assisted ventilation makes the end-expiratory oxygen concentration (EtO2) > 90%, wear the HFNO device according to the pre-adjusted mode (temperature 34°C, oxygen concentration 100%, flow rate 50 litres per minute). The nasal cannula will remain in place until intubation is complete (including DLT intubation, direct FOB guidance, and DLT alignment with FOB). After securing the HFNO device, the glottis was exposed using a laryngoscope, and the DLT main tracheal cuff was passed through the glottis and paused under direct vision. Insert the DLT into the bronchial tube lumen of the DLT using the FOB, and then advance the DLT into the corresponding main bronchus under the guidance of the FOB. After confirming the appropriate depth of the catheter using the FOB, insert the DLT into the anesthesia machine to complete the intubation process. After the DLT was connected to the anesthesia machine and mechanical ventilation was started, the HFNO device was removed.
  Other Names: high flow nasal oxygen therapy
  Arms: HFNO group

SUMMARY:
With the continuous strengthening of the concept of rapid rehabilitation, great progress has been made in minimally invasive thoracic surgery, and thoracoscopic surgery has developed rapidly. Double-lumen endotracheal(DLT) intubation is still the most reliable way of intubation in lung surgery. However, hypoxemia faced during double-lumen intubation still threatens the perioperative safety of thoracic surgery patients. In recent years, high-flow nasal oxygenation (HFNO) has great potential in the field of anesthesia, especially playing a new and important role in the prevention and treatment of short-term hypoxia and life-threatening airway emergencies. However, the use of HFNO in pulmonary surgery patients with poor pulmonary function lacks evidence-based basis, and there are few reliable clinical data.

This study adopted a prospective, randomized, controlled, single-blind design. A total of 100 patients aged 18-60 years who underwent elective thoracoscopy-assisted pulmonary surgery were included and randomly divided into the experimental group: HFNO was used in the process of double-lumen intubation asphyxia; the control group: according to the traditional intubation process, No oxygen therapy equipment was used during intubation asphyxiation. The lowest blood oxygen saturation during intubation, the incidence of hypoxemia during intubation, perioperative complications, and postoperative hospital stay were compared between the two groups.

This study explores the advantages of HFNO in complex endotracheal intubation, assuming that HFNO can improve the oxygen saturation of double-lumen intubation; optimize the intubation method of DLT, and tap its new potential to prevent and manage emergency airway crisis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60;
* Patients planning to undergo video-assisted thoracoscopic (VATS) lung surgery requiring DLT intubation;
* Patients who agreed to participate in this study.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification > IV;
* Patients with severe nasal obstruction; expected difficult intubation or difficulty with mask ventilation;
* Morbid obesity [Body Mass Index (BMI)>35kg/m2)];
* Airway anatomical abnormalities;
* Abnormal coagulation function;
* Emergency surgery;
* Patients at high risk of reflux aspiration, including ileus, full stomach, esophageal reflux disease;
* Pregnant or breastfeeding women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Minimum blood oxygen saturation (SpO2) | After the DLT intubation
  Minimum SpO2 measured by capillary oximeter during DLT intubation. SpO2 was continuously monitored by the monitor every 1 second and recorded every 5 seconds, and the lowest SpO2 was recorded through the monitor by the recording personnel who were not involved in anesthesia management.

SECONDARY OUTCOMES:
The incidence of lowest SpO2<90% | After the DLT intubation
  Minimum SpO2 measured by capillary oximeter during DLT intubation. SpO2 was continuously monitored by the monitor every 1 second and recorded every 5 seconds, and the lowest SpO2 was recorded through the monitor by the recording personnel who were not involved in anesthesia management.
The incidence of lowest SpO2<95% | After the DLT intubation
  Minimum SpO2 measured by capillary oximeter during DLT intubation. SpO2 was continuously monitored by the monitor every 1 second and recorded every 5 seconds, and the lowest SpO2 was recorded through the monitor by the recording personnel who were not involved in anesthesia management.
DLT intubation time | After the DLT intubation
  The DLT intubation period was defined as: from the time the video laryngoscope was placed in the oral cavity, to the confirmation of the correct position of the DLT by the FOB, and the end of the insertion of the anesthesia machine.
End-tidal carbon dioxide partial pressure after intubation | After the DLT intubation
  When the tracheal intubation is completed, the monitor displays the partial pressure of carbon dioxide at the end of the first mechanical ventilation.
End-tidal oxygen concentration after intubation | After the DLT intubation
  When the tracheal intubation is completed, the monitor displays the end-expiratory oxygen concentration of the first mechanical ventilation.
The incidence of difficult airway | After the DLT intubation
  Difficult airway was defined as failure of videolaryngoscope intubation, switch to fiberoptic bronchoscope-guided intubation.
The incidence of bronchial dislocation | After the DLT intubation
  Left or right bronchial tube strayed into right or left bronchus.
Incidence of related complications during intubation | After the DLT intubation
  Associated complications during intubation include: reflux aspiration, laryngospasm or bronchospasm, tracheal or bronchial tear, barotrauma, systolic blood pressure < 90 mmHg or initiation of vasoactive drugs, systolic blood pressure > 180 mmHg, severe arrhythmias, and lips or tooth damage.
Operator satisfaction with intubation | After the DLT intubation
  Operator satisfaction rating for intubation (range 0-10, with 0 being very dissatisfied and 10 being very satisfied).
The incidence of low blood oxygen saturation (SpO2<90%) in the post-anaesthesia care unit (PACU) | Up to 1 week
  After the patient entered the PACU, the blood oxygen saturation was continuously monitored and the lowest blood oxygen saturation value was recorded.
The incidence of postoperative airway-related complications | 1st, 2nd and 3rd day after surgery
  Postoperative airway-related complications include: sore throat, hoarseness, and nasopharyngeal dryness.
The incidence of nausea and vomiting | 1st, 2nd and 3rd day after surgery
  Interview patients' subjective feelings, including nausea and vomiting.
Patient satisfaction with anesthesia | The first day after surgery
  Patient satisfaction with anesthesia(range 0-10, with 0 being very dissatisfied and 10 being very satisfied).
Postoperative hospital stay | Through study completion, an average of 4 weeks
  The medical record system queries the number of days in hospital after surgery.
The incidence of postoperative complication | Through study completion, an average of 4 weeks
  Postoperative complications included postoperative atelectasis, pneumothorax, pulmonary infection, pleural effusion, bronchopleural fistula and postoperative bleeding.

IPD SHARING:
Plan to Share IPD: No
The research protocol will be announced later in the plan.

REFERENCES:
- [Background] Law JA, Duggan LV, Asselin M, Baker P, Crosby E, Downey A, Hung OR, Kovacs G, Lemay F, Noppens R, Parotto M, Preston R, Sowers N, Sparrow K, Turkstra TP, Wong DT, Jones PM; Canadian Airway Focus Group. Canadian Airway Focus Group updated consensus-based recommendations for management of the difficult airway: part 2. Planning and implementing safe management of the patient with an anticipated difficult airway. Can J Anaesth. 2021 Sep;68(9):1405-1436. doi: 10.1007/s12630-021-02008-z. Epub 2021 Jun 8. PMID 34105065
- [Background] Spence EA, Rajaleelan W, Wong J, Chung F, Wong DT. The Effectiveness of High-Flow Nasal Oxygen During the Intraoperative Period: A Systematic Review and Meta-analysis. Anesth Analg. 2020 Oct;131(4):1102-1110. doi: 10.1213/ANE.0000000000005073. PMID 32925331
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Kim HJ, Asai T. High-flow nasal oxygenation for anesthetic management. Korean J Anesthesiol. 2019 Dec;72(6):527-547. doi: 10.4097/kja.19174. Epub 2019 Jun 5. PMID 31163107
- [Background] Renda T, Corrado A, Iskandar G, Pelaia G, Abdalla K, Navalesi P. High-flow nasal oxygen therapy in intensive care and anaesthesia. Br J Anaesth. 2018 Jan;120(1):18-27. doi: 10.1016/j.bja.2017.11.010. Epub 2017 Nov 21. PMID 29397127
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Fong KM, Au SY, Ng GWY. Preoxygenation before intubation in adult patients with acute hypoxemic respiratory failure: a network meta-analysis of randomized trials. Crit Care. 2019 Sep 18;23(1):319. doi: 10.1186/s13054-019-2596-1. PMID 31533792
- [Derived] He R, Fang Y, Jiang Y, Yao D, Li Z, Zheng W, Liu Z, Luo N. High-flow nasal oxygenation versus face mask oxygenation for preoxygenation in patients undergoing double-lumen endobronchial intubation: protocol of a randomised controlled trial. BMJ Open. 2024 Mar 14;14(3):e080422. doi: 10.1136/bmjopen-2023-080422. PMID 38485472